CLINICAL TRIAL: NCT02212951
Title: A Single-blind Crossover Study of the Pharmacokinetic and Postprandial Glucose Dynamics of BIOD-531 Compared to Humulin R U-500 and Humalog Mix 75/25 in Subjects With Type 2 Diabetes Mellitus Who Are Treated With 50-200 Units of Insulin Per Day
Brief Title: Comparison of Postprandial Glucose Control Associated With BIOD-531 vs. Humalog Mix 75/25 vs. Humulin R U-500
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 3-152
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIOD-531 pre-meal (Experimental): Subcutaneous injection of 0.6 U/kg immediately before the start of the standardized breakfast
  Interventions: Drug: BIOD-531
- Humalog Mix 75/25 pre-meal (Active Comparator): Subcutaneous injection of 0.6 U/kg immediately before the start of the standardized breakfast
  Interventions: Drug: Humalog Mix 75/25
- Humulin R U-500 (Active Comparator): Subcutaneous injection of 0.6 U/kg immediately before the start of a standardized breakfast
  Interventions: Drug: Humulin R U-500
- BIOD-531 post-meal (Experimental): Subcutaneous injection of 0.6 U/kg 20 minutes after the start of the standardized breakfast
  Interventions: Drug: BIOD-531

INTERVENTIONS:
Drug: BIOD-531
  Arms: BIOD-531 post-meal; BIOD-531 pre-meal
Drug: Humalog Mix 75/25
  Arms: Humalog Mix 75/25 pre-meal
Drug: Humulin R U-500
  Arms: Humulin R U-500

SUMMARY:
The study is to compare meal time glucose control associated with BIOD-531, a rapidly absorbed concentrated insulin to that associated with Humalog Mix 75/25 and Humulin R U-500.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* BMI > 25 kg/m2
* Type 2 Diabetes Mellitus
* HbA1c < 10.0%
* Subject uses 50-200 units of insulin/day

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* History of bariatric surgery
* Corticosteroid therapy
* Significant cardiovascular or other major organ disease
* Females who are breast feeding or pregnant
* A sexually active person not using adequate contraceptive methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Post-standardized meal glucose exposure (AUC) | 0-120 minutes after meal

SECONDARY OUTCOMES:
Speed of insulin absorption (Times to 50%, 90%, maximal insulin concentrations) | 0-720 minutes
Insulin exposure (AUC) | Various time frames over 720 minutes
Maximal insulin concentration | 0-720 minutes
Post breakfast and post-lunch glucose exposure (AUC) | Various times frames over 720 minutes
Post-breakfast and post-lunch maximal glucose concentrations | 0-720 minutes
Injection site toleration (VAS and severity scales) | 30 minutes post injection
Draize injection site erythema and edema scoring | 0-720 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States